CLINICAL TRIAL: NCT06039111
Title: Indocyanine Green for Detection of Sentinel Lymph Nodes In Comparison to ICG Plus Technetium in the Evaluation of Vulvar Squamous Cell Carcinoma: The IGNITE-V Study
Brief Title: Indocyanine Green for Detection of Sentinel Lymph Nodes In Comparison to ICG Plus Technetium in the Evaluation of Vulvar Squamous Cell Carcinoma
Acronym: IGNITE-V
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Juravinski Cancer Centre Foundation (Other)
Responsible Party: Principal Investigator, Andra Nica, Gynecologic Oncologist, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16315
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Vulvar Cancer
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Sequential ICG and Technetium Detection (Experimental)
  Interventions: Procedure: ICG alone

INTERVENTIONS:
Procedure: ICG alone — SLNs will be detected with ICG alone, labelled as such, and subsequent to that tested with Gamma probe for accuracy

SUMMARY:
The aim of this study is to confirm prospectively if the use of near infrared-indocyanine green (NIR-ICG) alone offers similar accuracy and sensitivity to the gold standard dual technique for sentinel lymph node detection in early stage vulvar cancer.

ELIGIBILITY:
Inclusion Criteria:

Adult women (18 years of age) with FIGO Stage IB (> 1 mm depth of invasion) and small Stage II (4 cm) vulvar squamous cell carcinoma or cutaneous melanoma who are candidates for the Sentinel lymph node technique will be included (Negative clinical groin examination and/or imaging and primary unifocal vulvar tumor size of < 4 cm).

Exclusion Criteria:

Women with a prior history of pelvic, vulvovaginal or inguinal radiation, with allergy or hypersensitivity to Technetium or ICG, or Bartholin gland cancer will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
false-negative rate of the detection technique using ICG alone compared to ICG and Technetium (Dual method) per groin | 2 years
  This will be calculated as the number of groins for which positive SLN were missed using ICG alone; i.e. the number of groins for which ICG did not detect a positive SLN but was detected by ICG and Technetium, divided by the number of groins for which surgery was performed.

SECONDARY OUTCOMES:
1. The proportion of positive SLN detected by ICG for each groin divided by the total number of positive SLN detected using ICG and Technetium. | 2 years
  the unit of analysis is the number of SLN for each groin.

OTHER OUTCOMES:
2. The proportion of groins for which all SLN extracted were identified by ICG. | 2 years
  This is defined as the number of groins for whom, all SLN extracted were identified by ICG compared to the number of SLN extracted by ICG and Technetium.
3. The proportion of SLN extracted by ICG for each groin divided by the total number of SLN extracted using ICG and Technetium. | 2 years
  The unit of analysis is the number of SLN for each groin.
4. Rate of successful mapping of at least 1 SLN (per groin) | 2 years
  proportion
5. The specificity of positive SLN detected and number of SLN extracted by ICG will also be calculated, looking at the number of SLN which were detected by ICG alone. | 2 years
  Appropriate caution will be performed when looking at this outcome, understanding that evaluation of whether Technetium detected a SLN will be performed after the SLN is extracted, which is not consistent with normal practice and could be subject to bias.

IPD SHARING:
Plan to Share IPD: Undecided